CLINICAL TRIAL: NCT03587675
Title: Validation Screening Protocol for the Diagnosis of Exercise-induced Bronchoconstriction in Young Elite Athletes (13-18 y)
Brief Title: Diagnosis of EIB in Young Elite Athletes (13-18 y)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S59778
Record Dates: First submitted 2018-06-19; First posted 2018-07-16 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Exercise Induced Bronchospasm; Athletes; Adolescent
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Patch Tests

STUDY DESIGN:
Intervention Model Description: adolescents from different athletic disciplines and recreational adolescents will be tested for atopy, exercise-induced bronchospasm measured by EVH and biomarkers for EIB will be studied in blood and induced sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVH in high-school elite athletes (Other): EVH-test, skin prick test, sputum induction in all subjects Interventional but no drug or device tested
  Interventions: Diagnostic Test: EVH test

INTERVENTIONS:
Diagnostic Test: EVH test
  Other Names: sputum induction; skin prick test; peripheral blood test; nasal lavage

SUMMARY:
The investigators recently observed airway inflammation and increased damage-associated molecular pattern (DAMP) level in sputum of children (age 11-12y) and adolescents (18-23y) from elite sport programs in Belgium with increased risk of bronchoconstriction upon extreme exercise. They here want to validate these findings in a cohort 13-18y.

DETAILED DESCRIPTION:
State of the art Physical exercise, though absolutely beneficial for human well-being, is a well-known trigger to induce bronchoconstriction. Aretaeus of Cappadocia described the first cases of asthma triggered by exercise, already in the second century AD. Exercise can provoke bronchoconstriction in subjects with pre-existing asthma but can also induce bronchoconstriction in otherwise healthy subjects. The latter phenomenon is called exercise-induced bronchoconstriction (EIB). EIB is frequent in the general population and might affect between 5 and 10% of them, although population based reports are scarce. EIB is most prevalent in individuals performing endurance sport disciplines, such as long distance running, duathlon and triathlon, cycling and cross-country skiing. Due to frequent intense physical training, its incidence is higher in elite athletes compared to non-elite athletes. Its prevalence in elite athletes within these endurance sport disciplines is estimated to be up to 13%. The percentage in aquatic endurance sports was surprisingly even higher and reached 20% in the Olympic games of 2008. Besides intense physical training, environmental factors such as chlorine or cold air exposure are therefore also linked to the appearance of EIB.

The mechanism of exercise-induced bronchoconstriction is not fully clear: airway cooling resulting from conditioning of inspired air and post-exercise rewarming of airways have been proposed as "thermal" mechanism. However, airway dehydration as a result of increased ventilation, resulting in "augmented osmolarity" of the airway-lining fluid, seems to be a major cause. This augmented osmolarity is thought to trigger the release of mediators, such as histamine, cysteinyl leukotrienes and prostaglandins, from airway inflammatory cells, which leads to airway smooth-muscle contraction and airway edema. Last but not least, recent evidence, including data from the investigator' s laboratory, points to "epithelial damage" due to the high ventilation rate, with subsequent release of epithelial cell mediators, as underlying mechanism. This damage, which can be more pronounced if additional triggers are present, might lead to uncontrolled airway inflammation, can exacerbate the process and increase exercise-induced bronchoconstriction, potentially leading to persistent asthma. It is suggested that airway inflammation differ between subjects/athletes with pre-existing asthma (in whom airway eosinophils and Th2 inflammation are present) and those with EIB that developed during their career (in whom neutrophils and Th17 inflammation are present). If symptoms develop during their career, a causal relationship between the intense exercise and EIB can easily be suspected. In order to determine the exact moment of EIB development during their career, longitudinal studies, starting before EIB is present, are needed. Indeed, most adolescent elite athletes start their intense training protocols long before they start to perform at the highest international level.

If diagnosing EIB in adult elite athletes is difficult, its diagnosis in elite high-school athletes is a terrible challenge. Indeed, different diagnostic tests have been suggested by the International Olympic Committee-Medical Commission (IOC-MC) to identify EIB in adult elite athletes. If upon symptoms, classical diagnosis of asthma (e.g. by performing reversibility test after Salbutamol® inhalation) is excluded, airway hyperresponsiveness should be documented with the use of bronchoprovocation testing. These tests include direct challenges (e.g., with inhaled methacholine), which act on airway smooth muscle to cause bronchoconstriction, and indirect challenges, such as Eucapnic Voluntary Hyperpnea (EVH) particularly recommended for athletes, hyperosmolar tests with saline or mannitol, and laboratory or field exercise tests. However, athletes may have a positive response (with a drop in Forced expiratory volume in one second (FEV1) above the cited cut-off) to only one of these types of tests. Therefore, more than one type of test may be needed, and ideally the testing should be performed during a period of intense training.

The investigators recently adapted the EVH test, gold standard diagnostic test recommended by IOC-MC to diagnose EIB in elite athletes for its use in teenagers. Instead of the maximal voluntary ventilation (MVV) of 85% during 6 minutes, usually requested in adult subjects (which is 30XFEV1, but would mean an unrealistic performance of 100% of MVV in adolescents), a ventilatory target of 70% which corresponds to 21 x FEV1 in young athletes is feasible for the majority of athletes (see table 1). Therefore the test aims at a ventilation target of 70% during 6 minutes. Moreover, to exclude exhaustion as a cause of artificial FEV1 drop, the change in Tiffeneau index (TI=FEV1/FVC) was also calculated. Only if TI at the time of maximal fall minus TI at baseline was below zero, the fall in FEV1 is thought to reflect true airway obstruction.

With those small adaptations, the test can be performed in almost all high-school elite athletes aged 12-14 years. Surprisingly, 23% percent of basketball players (3/13), 21% of football players (4/19) and up to 54% of swimmers (6/11) aged 12-14 years, had a positive EVH test at enrollment to an elite sport program compared to 13% of control subjects. During the longitudinal observation (registered at clinicaltrials.gov (NCT02432183) unpublished results), two out of four football players with a positive EVH test, terminated their high-school elite program early. Although sport technical reasons might also be the limiting factor to continue the program, their EIB can also explain impaired performance that can ensue if preventive measures are not taken. It is however not yet clear which medical treatment ideally should be used in those elite athletes. Nevertheless, several treatment opportunities exist, which might at least enable them to perform their sports in optimal conditions.

Performing EVH tests as a screening test yearly in all high-school athletes is labor-extensive and at high cost. The investigators therefore studied whether questionnaires might help to indicate young (12-14 years) athletes at risk to have a positive EVH test. They were able to test the validated AQUA (Allergy Questionnaire for Athletes) Questionnaire for adults and adolescents, in a young elite athletes cohort. By performing skin prick tests in those subjects to search for allergy, if the AQUA score was ≥ 5, the test predicted atopy with a specificity of 78% and a sensitivity of 62.5%

% Of MVV Adults Adolescents (12-14 y) 100% 35 × FEV1 30 × FEV1 85% 30 × FEV1 70% 21 × FEV1 60% 21 × FEV1

Table 1 Comparison of maximal ventilatory capacity between adults and adolescents

The investigators found that atopic individuals in the cohort had increased risk to test positive for EIB (Fisher exact test p=0.04). However, due to the high number of subjects with a positive EIB test but negative AQUA questionnaire, the AQUA questionnaire by itself can't be used to predict EIB (p=0.4). However, one out of five questions added by our group to this questionnaire ("Do you suffer from wheeze during exercise?") by itself predicted EIB with 93% specificity and 24% sensitivity. Adding a second question to this ("Has a doctor ever diagnosed you with an allergic condition?") increased the specificity to predict a positive EIB test to 99% but lowered sensitivity to 15% only (manuscript in preparation).

Question 1 Do you suffer from wheeze during exercise ? Question 2 Do you experience shortness of breath during exercise? Question 3 Has a doctor ever diagnosed you with an allergic condition? Question 4 Do you frequently suffer from upper respiratory tract infections or fever? Question 5 Is anyone in your family allergic?

Table 2. Questions added to AQUA questionnaire in screening protocol of 12-14y high-school elite athletes

These findings formed basis for the current idea about how to screen for EIB in young elite athletes A/ If the young athlete answers positive to question 1, "Do you suffer from wheeze during exercise ?", A.1 asthma has to be excluded (by Salbutamol reversibility test) A.2 EIB can be searched for by EVH test. B/ If the child has a positive AQUA score (>5), B.1. atopy might be present and can be searched for by CAPtest and/or SPT. B.1.a If atopy tests are positive, EIB can be tested by EVH test. B.1.b If atopy tests are negative, a watch-full waiting strategy can be chosen

Those questionnaires can easily be repeated yearly

However, although this would be a great advantage in the screening process of young athletes, this pilot study should at least be repeated in an older age group of athletes (13-18 years). Moreover, the question still remains whether we need to perform different tests to diagnose EIB and whether a hierarchical structure in those tests can be chosen. Indeed, in daily routine, EVH test at the UZ Leuven is restricted for those subjects in whom histamine provocation test is negative but EIB is highly suspected, based on clinical history. It is not known whether all subjects with positive histamine provocation test also have positive EIB.

Finally, sputum IL-1beta-low subjects, in the absence of atopy, had a very low chance to have positive EVH testing (Fisher exact test p=0.0088; compared to 0.04 for atopy alone, see higher). Adding sputum cytokine IL-1beta mRNA detection to the screening protocol might therefore increase the negative predictive value of the flow chart. However, performing induced sputum is also challenging and cytokine mRNA detection in the samples (though routinely performed in the investigator's laboratory) is still no routine procedure.

Hypotheses The investigators hypothesize that the findings in the first young cohort will be similar or even more pronounced in the slightly older cohort of athletes. This means that

1. they hypothesize that AQUA questionnaire can also predict atopy in this age group
2. they hypothesize that atopy will be a risk factor for EIB in that age group
3. they consider EVH test (in the absence of asthma) to be the best test to detect EIB (in comparison to histamine provocation test) in that age group
4. they hypothesize that a positive AQUA score and/or a positive score to question 1 and 3 of table 2 can be used to screen for EIB (as outlined in figure 2)
5. they hypothesize that adding sputum cytokine mRNA detection might increase the negative predictive value of the screening protocol

Aim of the study Therefore the aim of the study is to study the existence of EIB in high school elite athletes as well as athletes performing at least 12 hours sport a week aged 13-18 years (n=50). More specifically the investigators want

1. to compare the proportion of EIB positive subjects (defined as ≥10% fall in FEV1 at least 5' after EVH provocation) between those athletes and age matched controls (n=20).
2. to correlate the answers in the questionnaires with the existence of EIB in the cohort
3. to correlate the PC20 (by histamine provocation test) with the % max fall in EVH test in the cohort
4. to study sputum mRNA levels in correlation to the presence of EIB in the cohort

Material and method

young athletes (swimmers, indoor and outdoor athletes) performing at least 12 hours sport a week and controls performing less than 6 hours sport a week will be recruited. To that aim, the investigators have a close collaboration with the Sport Medical Advice Center (SMAC UZ Leuven) screening all high-school elite athletes from 'topsportschool' Leuven, as well as with the medical coordinators of the Flemish Swimming Federation, Basketball federation and Football federation. Controls will be recruited amongst children and relatives from personnel.

Questionnaires (AQUA and table 2), skin prick tests for common environmental allergens, venous puncture, sputum induction, reversibility test after Salbutamol inhalation, FENO measurement, histamine provocation test, EVH test and/or exercise field test will be performed in these subjects.

Specific IgE to allergens will be measured by CAPtest. Biomarkers such as serum CC16 will be measured by ELISA. Sputum differential cell count will be done by cytospin and cytokine mRNA detection by RT-PCR. Merocell obtained nasal lavage fluid biomarkers will be studied by ELISA. All tests together will take +/-1.30h. If trainers from a specific discipline consider this too busy, we can omit one or more of the following: sputum induction, Merocell and/or skin prick tests. In case of the latter, allergy diagnosis will be based on CAPtest only. This will be discussed in advance with trainers and sport doctors and manually added to the IC/assent documents, if this is the case.

Spirometry, EVH test and histamine provocation test are routinely performed in the hospital.

Statistical analysis Sample size calculation has not been done, as all Flemish elite high-school athletes within the cited sport disciplines (which are the largest branches in B) will be invited. Prior studies revealed that more than 95% of them are willing to participate. Based on the results of the previous study in the younger age group in an even smaller sample size, the investigators consider the current sample size sufficient for this study.

1. Fisher exact test (or Chi-square in case of the different disciplines separately) will be used to study whether the proportion of athletes with positive EVH test (at the cited cut-off) is significantly different from its proportion in healthy subjects
2. Differences in absolute maximal fall in FEV1, serum biomarkers, specific sputum cytokine mRNA levels and sputum cellular counts between athletes and controls after EVH provocation will be studied by two-tailed (one-tailed where appropriate) non-parametric Mann-Whitney-U test (or if normality test is passed, by parametric t test). Differences amongst the sports branches will be studied by Kruskall-Wallis (or ANOVA if normality test is passed) with adequate post-tests.
3. Sensitivity, specificity, PPV and NPV (as well as ROC curves) to study the usefulness of the AQUA questionnaire and/or the cited 5 questions and/or IL-1beta-low sputum mRNA levels, to predict atopy on the one hand and positive EVH test on the other hand, will be calculated.
4. Correlation between PC20 and max fall in FEV will be studied by Spearman correlation test without or with prior data (e.g. log) transformation.

Statistical analysis will be performed by Prism Graph 7

Expected result

The investigators expect to be able to repeat the findings observed in the younger age groups. Moreover, they expect to be able to increase sensitivity of the screening protocol and increase the negative predictive value of the screening test. To that latter aim, sputum IL-1beta mRNA measurement might be of help.

Potential risk

Because only a limited group of 13-18 year old athletes (n=50) is studied, the study might lack power to obtain the goal. Power analysis has not been performed, as the study is limited by the number of elite high-school students in the 'topsportschool'.

Feasibility

FWO-TBM study granted

ELIGIBILITY:
Inclusion Criteria:

* high-school elite athletes from 'topsportschool' or 'future team'
* from following disciplines: swimming, basket, volley or foot ball
* performing at least 12 h sport a week

or

* healthy recreational control subjects
* performing less than 6 hours sport/week

Exclusion Criteria:

- acute infection in four weeks prior to test

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
incidence of athletes with exercise-induced bronchospasm | 2 years
  measured by positive EVH test: at least 10% drop in FEV1% between 5-20' after EVH

SECONDARY OUTCOMES:
use of questionnaire to predict positive EVH test | 2 years
  AQUA questionnaire+additive questions (n=5)
use of blood biomarker to predict positive EVH test | 3 years
  blood CC16 levels measured by ELISA
use of sputum biomarker to predict negative EVH test | 3 years
  sputum IL-1 beta mRNA levels measured by q-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MA Bullens, MD, PhD, Principal Investigator — Lab pediatric Immunology, Dep Microbiology and Immunology
Locations (1):
- University Hospital of Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
Plan from KU Leuven will be followed

REFERENCES:
- [Background] Carlsen KH, Carlsen KC. Exercise-induced asthma. Paediatr Respir Rev. 2002 Jun;3(2):154-60. PMID 12297065
- [Background] Boulet LP, O'Byrne PM. Asthma and exercise-induced bronchoconstriction in athletes. N Engl J Med. 2015 Feb 12;372(7):641-8. doi: 10.1056/NEJMra1407552. No abstract available. PMID 25671256
- [Background] Fitch KD, Sue-Chu M, Anderson SD, Boulet LP, Hancox RJ, McKenzie DC, Backer V, Rundell KW, Alonso JM, Kippelen P, Cummiskey JM, Garnier A, Ljungqvist A. Asthma and the elite athlete: summary of the International Olympic Committee's consensus conference, Lausanne, Switzerland, January 22-24, 2008. J Allergy Clin Immunol. 2008 Aug;122(2):254-60, 260.e1-7. doi: 10.1016/j.jaci.2008.07.003. PMID 18678340
- [Background] Mountjoy M, Fitch K, Boulet LP, Bougault V, van Mechelen W, Verhagen E. Prevalence and characteristics of asthma in the aquatic disciplines. J Allergy Clin Immunol. 2015 Sep;136(3):588-94. doi: 10.1016/j.jaci.2015.01.041. Epub 2015 Mar 24. PMID 25819982
- [Background] Hallstrand TS, Moody MW, Wurfel MM, Schwartz LB, Henderson WR Jr, Aitken ML. Inflammatory basis of exercise-induced bronchoconstriction. Am J Respir Crit Care Med. 2005 Sep 15;172(6):679-86. doi: 10.1164/rccm.200412-1667OC. Epub 2005 Jun 9. PMID 15947280
- [Background] Anderson SD, Kippelen P. Airway injury as a mechanism for exercise-induced bronchoconstriction in elite athletes. J Allergy Clin Immunol. 2008 Aug;122(2):225-35; quiz 236-7. doi: 10.1016/j.jaci.2008.05.001. Epub 2008 Jun 12. PMID 18554705
- [Background] Helenius I, Lumme A, Haahtela T. Asthma, airway inflammation and treatment in elite athletes. Sports Med. 2005;35(7):565-74. doi: 10.2165/00007256-200535070-00002. PMID 16026170
- [Background] Perry C, Pick M, Bdolach N, Hazan-Halevi I, Kay S, Berr I, Reches A, Harishanu Y, Grisaru D. Endurance exercise diverts the balance between Th17 cells and regulatory T cells. PLoS One. 2013 Oct 9;8(10):e74722. doi: 10.1371/journal.pone.0074722. eCollection 2013. PMID 24130669
- [Background] Rundell KW, Slee JB. Exercise and other indirect challenges to demonstrate asthma or exercise-induced bronchoconstriction in athletes. J Allergy Clin Immunol. 2008 Aug;122(2):238-46; quiz 247-8. doi: 10.1016/j.jaci.2008.06.014. PMID 18678339
- [Background] Chateaubriand do Nascimento Silva Filho MJ, Goncalves AV, Tavares Viana M, Peixoto DM, Cavalcanti Sarinho ES, Rizzo JA. Exercise-induced bronchoconstriction diagnosis in asthmatic children: comparison of treadmill running and eucapnic voluntary hyperventilation challenges. Ann Allergy Asthma Immunol. 2015 Oct;115(4):277-81. doi: 10.1016/j.anai.2015.07.009. Epub 2015 Aug 1. PMID 26238422
- [Background] Anderson SD, Argyros GJ, Magnussen H, Holzer K. Provocation by eucapnic voluntary hyperpnoea to identify exercise induced bronchoconstriction. Br J Sports Med. 2001 Oct;35(5):344-7. doi: 10.1136/bjsm.35.5.344. PMID 11579071
- [Background] Castricum A, Holzer K, Brukner P, Irving L. The role of the bronchial provocation challenge tests in the diagnosis of exercise-induced bronchoconstriction in elite swimmers. Br J Sports Med. 2010 Aug;44(10):736-40. doi: 10.1136/bjsm.2008.051169. Epub 2008 Oct 23. PMID 18948353
- [Background] Hull JH, Ansley L, Price OJ, Dickinson JW, Bonini M. Eucapnic Voluntary Hyperpnea: Gold Standard for Diagnosing Exercise-Induced Bronchoconstriction in Athletes? Sports Med. 2016 Aug;46(8):1083-93. doi: 10.1007/s40279-016-0491-3. PMID 27007599
- [Background] Bonini M, Braido F, Baiardini I, Del Giacco S, Gramiccioni C, Manara M, Tagliapietra G, Scardigno A, Sargentini V, Brozzi M, Rasi G, Bonini S. AQUA: Allergy Questionnaire for Athletes. Development and validation. Med Sci Sports Exerc. 2009 May;41(5):1034-41. doi: 10.1249/MSS.0b013e318193c663. PMID 19346984
- [Background] Truyen E, Coteur L, Dilissen E, Overbergh L, Dupont LJ, Ceuppens JL, Bullens DM. Evaluation of airway inflammation by quantitative Th1/Th2 cytokine mRNA measurement in sputum of asthma patients. Thorax. 2006 Mar;61(3):202-8. doi: 10.1136/thx.2005.052399. Epub 2006 Jan 31. PMID 16449261
- [Background] Bullens DM, Truyen E, Coteur L, Dilissen E, Hellings PW, Dupont LJ, Ceuppens JL. IL-17 mRNA in sputum of asthmatic patients: linking T cell driven inflammation and granulocytic influx? Respir Res. 2006 Nov 3;7(1):135. doi: 10.1186/1465-9921-7-135. PMID 17083726
- [Background] Bullens DM, Decraene A, Dilissen E, Meyts I, De Boeck K, Dupont LJ, Ceuppens JL. Type III IFN-lambda mRNA expression in sputum of adult and school-aged asthmatics. Clin Exp Allergy. 2008 Sep;38(9):1459-67. doi: 10.1111/j.1365-2222.2008.03045.x. Epub 2008 Jun 28. PMID 18564328
- [Background] Grabowski M, Kasran A, Seys S, Pauwels A, Medrala W, Dupont L, Panaszek B, Bullens D. Pepsin and bile acids in induced sputum of chronic cough patients. Respir Med. 2011 Aug;105(8):1257-61. doi: 10.1016/j.rmed.2011.04.015. Epub 2011 May 17. PMID 21592756
- [Background] Bobic S, Seys S, De Vooght V, Callebaut I, Hox V, Dooms C, Vinckier S, Jonckx B, Saint-Remy JM, Stassen JM, Bullens DM, Ceuppens JL, Carmeliet P, Hellings PW. Placental growth factor contributes to bronchial neutrophilic inflammation and edema in allergic asthma. Am J Respir Cell Mol Biol. 2012 Jun;46(6):781-9. doi: 10.1165/rcmb.2011-0152OC. Epub 2012 Jan 20. PMID 22268141
- [Background] Grabowski M, Seys S, Decraene A, Kasran A, Dilissen E, Barg W, Medrala W, Dupont LJ, Panaszek B, Bullens DM. Airway inflammation in patients with chronic non-asthmatic cough. Thorax. 2013 Feb;68(2):125-30. doi: 10.1136/thoraxjnl-2012-201895. Epub 2012 Oct 23. PMID 23093651
- [Background] Seys SF, Grabowski M, Adriaensen W, Decraene A, Dilissen E, Vanoirbeek JA, Dupont LJ, Ceuppens JL, Bullens DM. Sputum cytokine mapping reveals an 'IL-5, IL-17A, IL-25-high' pattern associated with poorly controlled asthma. Clin Exp Allergy. 2013 Sep;43(9):1009-17. doi: 10.1111/cea.12125. PMID 23957336
- [Background] Marijsse GS, Seys SF, Schelpe AS, Dilissen E, Goeminne P, Dupont LJ, Ceuppens JL, Bullens DM. Obese individuals with asthma preferentially have a high IL-5/IL-17A/IL-25 sputum inflammatory pattern. Am J Respir Crit Care Med. 2014 May 15;189(10):1284-5. doi: 10.1164/rccm.201311-2011LE. No abstract available. PMID 24832749
- [Background] Steelant B, Hox V, Van Gerven L, Dilissen E, Dekimpe E, Kasran A, Aertgeerts S, Van Belle V, Peers K, Dupont LJ, Hellings PW, Bullens DM, Seys SF. Nasal symptoms, epithelial injury and neurogenic inflammation in elite swimmers. Rhinology. 2018 Sep 1;56(3):279-287. doi: 10.4193/Rhin17.167. PMID 29561921
- [Result] Seys SF, Hox V, Van Gerven L, Dilissen E, Marijsse G, Peeters E, Dekimpe E, Kasran A, Aertgeerts S, Troosters T, Vanbelle V, Peers K, Ceuppens JL, Hellings PW, Dupont LJ, Bullens DM. Damage-associated molecular pattern and innate cytokine release in the airways of competitive swimmers. Allergy. 2015 Feb;70(2):187-94. doi: 10.1111/all.12540. PMID 25358760
- [Result] Van der Eycken S, Schelpe A, Marijsse G, Dilissen E, Troosters T, Vanbelle V, Aertgeerts S, Dupont LJ, Peers K, Bullens DM, Seys SF. Feasibility to apply eucapnic voluntary hyperventilation in young elite athletes. Respir Med. 2016 Feb;111:91-3. doi: 10.1016/j.rmed.2015.12.012. Epub 2016 Jan 4. PMID 26790574
- [Result] Jonckheere AC, Seys SF, Dilissen E, Marijsse G, Schelpe AS, Van der Eycken S, Verhalle T, Vanbelle V, Aertgeerts S, Troosters T, Peers K, Dupont LJ, Bullens DMA. AQUA(c) Questionnaire as prediction tool for atopy in young elite athletes. Pediatr Allergy Immunol. 2018 Sep;29(6):648-650. doi: 10.1111/pai.12949. Epub 2018 Jul 9. No abstract available. PMID 29908073
- [Derived] Goossens J, Jonckheere AC, Seys SF, Dilissen E, Decaesteker T, Goossens C, Peers K, Vanbelle V, Stappers J, Aertgeerts S, De Wilde B, Leus J, Verelst S, Raes M, Dupont L, Bullens DM. Activation of epithelial and inflammatory pathways in adolescent elite athletes exposed to intense exercise and air pollution. Thorax. 2023 Aug;78(8):775-783. doi: 10.1136/thorax-2022-219651. Epub 2023 Mar 16. PMID 36927754